CLINICAL TRIAL: NCT03107104
Title: Topcon DRI OCT Triton (Plus) Fundus Autofluorescence and Fluorescein Angiography Image Quality Evaluation Study
Brief Title: Triton Fundus Autofluorescence and Fluorescein Angiography
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Triton FA FAF
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Medical Need for Fluorescein Angiography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Medical need for FA imaging: Subjects deemed to have a medical need for FA imaging will be imaged on the Topcon DRI OCT Triton (plus) and TRC-50DX retinal camera
  Interventions: Device: Topcon DRI OCT Triton (plus); Device: TRC-50DX retinal camera

INTERVENTIONS:
Device: Topcon DRI OCT Triton (plus) — The Topcon DRI OCT Triton (plus) is an OCT with a fundus camera used for diagnostic purposes
Device: TRC-50DX retinal camera — The TRC-50DX retinal camera is a fundus camera used for diagnostic purposes

SUMMARY:
Compare the image quality of the fundus autofluorescence and fluorescein angiography

DETAILED DESCRIPTION:
The objectives of this study are to:

1. Compare the image quality of the fundus autofluorescence (FAF) photographs between DRI OCT Triton (plus) and TRC-50DX retinal camera.
2. Compare the image quality of the fluorescein angiography (FA) photographs between DRI OCT Triton (plus) and TRC-50DX retinal camera.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be at least 18 years of age
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects who consent to, via clinic's standard FA consent form, and will undergo dye injection for FA imaging at the clinic visit based on medical need

Exclusion Criteria

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects with ocular media not sufficiently clear to obtain acceptable fundus images
3. Patients with ocular motility dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with medical need for FA imaging
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Fundus autofluorescence image quality | 1 Minute
  Comparison of DRI OCT Triton (plus) and TRC-50DX photographs
Fluorescein angiography image quality at 120 seconds to 300 seconds after dye injection | 120 seconds to 300 seconds
  Comparison of DRI OCT Triton (plus) and TRC-50DX photographs
Fluorescein angiography image quality at greater than 300 seconds after dye injection | greater than 300 seconds
  Comparison of DRI OCT Triton (plus) and TRC-50DX photographs

CONTACTS AND LOCATIONS:
Overall Officials: Charles Riesman, MS, Study Chair — Topcon Corporation
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No